CLINICAL TRIAL: NCT07216781
Title: Evaluating the Safety and Efficacy of Injectable Klotho Plasmid Gene Therapy in Humans: An Interventional, Non-Placebo-Controlled Pilot Phase Study
Brief Title: Safety and Efficacy of Injectable Klotho Plasmid Gene Therapy in Humans
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Minicircle (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MINICIRCLE-KLO
Record Dates: First submitted 2025-09-30; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adults
Keywords: Klotho; plasmid; gene therapy

STUDY DESIGN:
Intervention Model Description: Non-placebo-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schedule of Administration and Sample Selection (Experimental): This arm includes cognitive and health battery at multiple intervals pre- and post-administration of Klotho
  Interventions: Genetic: Injectable Plasmid Klotho Gene Therapy

INTERVENTIONS:
Genetic: Injectable Plasmid Klotho Gene Therapy — Injection of plasmid-delivered Klotho gene therapy

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of a gene therapy for Klotho, delivered via a nonviral plasmid in healthy adult volunteers. Additionally, this study seeks to understand the cognitive and health benefits of the Klotho gene therapy.

DETAILED DESCRIPTION:
Note that the investigational product will be administered at a site outside of the U.S. which is not under FDA jurisdiction, and only non-treatment pre/post outcome assessments (e.g., cognitive assessments or blood sample collection) occur at the U.S. site.

Participants will take part in cognitive and health testing before and after administration of plasmid-delivered Klotho gene therapy. The method of administration will be subcutaneous injection into abdominal fat deposits. Klotho may improve cognitive function, kidney function, healthspan, and lifespan. Healthy volunteers will partake in a series of blood draws, health screenings, questionnaires, brain perfusion/function measures, and cognitive testing multiple times before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participant is open to morphological change
* If female, participant agrees to maintain contraception
* If female, participant agrees to take a pregnancy test
* If female, participant agrees to a pregnancy waiver

Exclusion Criteria:

* Women of childbearing potential who are unwilling or unable to use effective contraception for the duration of the study
* History of cancer diagnosis
* Preexisting medical issues that may be exacerbated by the treatment
* Has received any gene therapy within the past 12 months
* Unwilling or unable to provide written informed consent

Ages: 23 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Concentration of Serum α-Klotho Measured by Enzyme-Linked Immunosorbent Assay (pg/mL) | Measured 1 month before and 7 days before injection, then 3 days, 7 days, 1 month, 3 months, 6 months after
  Serum α-Klotho protein concentration will be quantified using a validated enzyme-linked immunosorbent assay (ELISA). Results will be reported as picograms per milliliter (pg/mL) for each participant at each time point. Higher or lower values have no inherent directionality and will be interpreted in study context.
Adverse Events: Number and Percentage of Participants Experiencing Treatment-Emergent Adverse Events as Assessed Patient-Reported Outcomes Version of Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Measured 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Assessed through a checklist version of the PRO-CTCAE with each symptom options being none, mild, moderate, or severe. Items will be scored with 0, 1, 2, 3 respectively. Item responses will be summarized as number and percentage of participants experiencing each adverse event by system/organ class. High scores indicate highest severity of symptoms and low scores indicate no symptoms.
Concentration of Serum Fibroblast Growth Factor 23 (FGF23) Measured by Enzyme-Linked Immunosorbent Assay (pg/mL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Fibroblast Growth Factor 23 (FGF23) concentration will be quantified in serum using a validated enzyme-linked immunosorbent assay (ELISA). Results will be expressed in picograms per milliliter (pg/mL) for each participant and time point. FGF23 is a downstream effector of α-Klotho signaling and reflects activity of the phosphate-vitamin D regulatory axis.
Concentration of Intact Parathyroid Hormone Measured by Two-Site Immunoassay (pg/mL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Intact Parathyroid Hormone (PTH) will be measured in serum using a two-site immunoassay that detects the full-length molecule. Results will be reported in picograms per milliliter (pg/mL) per participant and time point. PTH reflects parathyroid activity within the α-Klotho-FGF23-vitamin D feedback pathway.
Concentration of Serum 1,25-Dihydroxyvitamin D (Calcitriol) Measured by Liquid Chromatography-Tandem Mass Spectrometry (pg/mL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum 1,25-dihydroxyvitamin D (calcitriol) will be quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS). Concentrations will be expressed in picograms per milliliter (pg/mL). This hormone regulates calcium and phosphate balance and is a downstream marker of α-Klotho-FGF23-PTH axis modulation.
Concentration of Serum Phosphorus Measured by Clinical Chemistry Analyzer (mg/dL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum inorganic phosphorus will be measured on a standard clinical chemistry analyzer. Results will be reported in milligrams per deciliter (mg/dL) for each participant and time point. Phosphorus levels reflect systemic phosphate homeostasis influenced by α-Klotho and FGF23 activity.
Urinary Phosphate Excretion Measured by Clinical Chemistry Assay (mg/24 h or mg/g Creatinine) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Urinary phosphate will be assessed using a validated chemistry assay. Results will be expressed either as total phosphate excretion in milligrams per 24 hours (mg/24 h) or as the phosphate-to-creatinine ratio (mg phosphate per g creatinine). This measure reflects renal handling of phosphate and functional effects of α-Klotho on phosphate excretion.
Concentration of Serum Cystatin C Measured by Immunoassay (mg/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum Cystatin C will be measured using a standardized immunoassay and reported in milligrams per liter (mg/L) for each participant and time point. Cystatin C serves as a biomarker of glomerular filtration rate and provides a mechanistic link between α-Klotho activity and renal function.

SECONDARY OUTCOMES:
Change From Baseline in World Health Organization Quality of Life Brief Version Domain Scores (0-100) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 month, 6 months after.
  The World Health Organization Quality of Life Brief Version (WHOQOL-BREF) is a self-report questionnaire that includes four domains: Physical Health, Psychological, Social Relationships, and Environment. Each domain score is transformed to a 0-100 scale, with higher scores indicating better quality of life. Changes from baseline will be reported for each domain separately.
Change From Baseline in Flanker Inhibitory Control and Attention Test T-Score (Mean 50 ± 10) | Measured 7 days before, then 3 days, 7 days, 1 month, 3 months, 6 months after treatment.
  The Flanker Inhibitory Control and Attention Test measures inhibitory control and attention. Scores are age-adjusted T-scores (mean 50, SD 10). Higher scores indicate better performance. Changes from baseline will be analyzed per participant and time point.
Change From Baseline in Dimensional Change Card Sort Test T-Score (Mean 50 ± 10) | Measured 7 days before, then 3 days, 7 days, 1 month, 3 months, 6 months after treatment.
  The Dimensional Change Card Sort Test assesses cognitive flexibility. Scores are age-adjusted T-scores (mean 50, SD 10). Higher scores indicate better executive function. Changes from baseline will be analyzed per participant and time point.
Change From Baseline in Pattern Comparison Processing Speed Test T-Score (Mean 50 ± 10) | Measured 7 days before, then 3 days, 7 days, 1 month, 3 months, 6 months after treatment.
  The Pattern Comparison Processing Speed Test measures processing speed using age-adjusted T-scores (mean 50, SD 10). Higher scores reflect faster cognitive processing. Changes from baseline will be analyzed per participant and time point.
Change From Baseline in Picture Sequence Memory Test T-Score, Forms A and B (Mean 50 ± 10) | Measured 7 days before, then 3 days, 7 days, 1 month, 3 months, 6 months after treatment.
  Picture Sequence Memory Test evaluates episodic memory. Each form (A and B) yields an age-adjusted T-score (mean 50, SD 10). Higher scores indicate better memory performance. Forms A and B will be averaged.
Change From Baseline in Picture Vocabulary Test T-Score (Mean 50 ± 10) | Measured 7 days before, then 3 days, 7 days, 1 month, 3 months, 6 months after treatment.
  Picture Vocabulary Test measures receptive vocabulary. Results are expressed as age-adjusted T-scores (mean 50, SD 10), with higher scores indicating better performance. Change from baseline will be analyzed per participant and time point.
Change From Baseline in Reynolds Intellectual Assessment Scales-Second Edition (RIAS-2) Composite Scores (Standard Score Mean 100 ± 15) | Measured 1 month before and then 1 month and 3 months after.
  The Reynolds Intellectual Assessment Scales-Second Edition (RIAS-2) measures verbal, nonverbal, and composite intelligence. Each index yields a standard score (mean 100, SD 15) and subtests yield scaled scores (mean 10, SD 3). Higher scores indicate better cognitive performance. Changes from baseline will be reported for each selected index separately.
Concentration of Serum Glucose Measured by Clinical Chemistry Analyzer (mg/dL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum glucose will be measured using a standard clinical chemistry analyzer and expressed in milligrams per deciliter (mg/dL). Elevated glucose may indicate altered carbohydrate metabolism or metabolic stress.
Concentration of Total Serum Calcium Measured by Clinical Chemistry Analyzer (mg/dL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Total calcium will be quantified using a colorimetric method on a clinical chemistry analyzer. Results will be expressed in milligrams per deciliter (mg/dL). Calcium levels reflect bone-mineral balance and parathyroid function.
Concentration of Ionized Calcium Measured by Ion-Selective Electrode (mmol/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Ionized calcium will be measured using an ion-selective electrode analyzer. Results will be reported in millimoles per liter (mmol/L) and represent physiologically active calcium fraction.
Concentration of Serum Sodium Measured by Ion-Selective Electrode (mmol/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Sodium concentration will be measured using an ion-selective electrode analyzer and expressed in millimoles per liter (mmol/L). Sodium reflects hydration and electrolyte balance.
Concentration of Serum Potassium Measured by Ion-Selective Electrode (mmol/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum potassium will be quantified using an ion-selective electrode analyzer and expressed in millimoles per liter (mmol/L). Potassium levels reflect renal and electrolyte homeostasis.
Concentration of Serum Chloride Measured by Ion-Selective Electrode (mmol/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum chloride will be measured using an ion-selective electrode analyzer. Results will be expressed in millimoles per liter (mmol/L) and reflect acid-base and hydration status.
Concentration of Serum Bicarbonate (CO₂) Measured by Clinical Chemistry Analyzer (mmol/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum bicarbonate will be measured as total CO₂ on a clinical chemistry analyzer. Results will be expressed in millimoles per liter (mmol/L) and indicate systemic acid-base balance.
Concentration of Blood Urea Nitrogen (BUN) Measured by Clinical Chemistry Analyzer (mg/dL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Blood urea nitrogen (BUN) will be measured using a standard enzymatic assay and expressed in milligrams per deciliter (mg/dL). BUN reflects renal function and nitrogen metabolism.
Concentration of Serum Creatinine Measured by Clinical Chemistry Analyzer (mg/dL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum creatinine will be measured using a validated enzymatic method on a clinical chemistry analyzer. Results will be reported in milligrams per deciliter (mg/dL) and serve as an indicator of renal filtration.
Concentration of Serum Albumin Measured by Clinical Chemistry Analyzer (g/dL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum albumin will be quantified using a bromocresol green dye-binding method and expressed in grams per deciliter (g/dL). Albumin reflects nutritional status and hepatic synthetic function.
Concentration of Total Serum Protein Measured by Biuret Method (g/dL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Total protein will be measured using the biuret colorimetric assay and expressed in grams per deciliter (g/dL). This parameter provides an overview of plasma protein balance.
Concentration of Alkaline Phosphatase (ALP) Measured by Clinical Chemistry Analyzer (IU/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum alkaline phosphatase will be quantified by an enzymatic colorimetric method and expressed in international units per liter (IU/L). ALP reflects hepatobiliary and bone function.
Concentration of Alanine Aminotransferase (ALT) Measured by Clinical Chemistry Analyzer (IU/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum ALT activity will be measured enzymatically and expressed in international units per liter (IU/L). ALT serves as a marker of hepatocellular injury.
Concentration of Aspartate Aminotransferase (AST) Measured by Clinical Chemistry Analyzer (IU/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Serum AST activity will be determined by an enzymatic method and expressed in international units per liter (IU/L). AST reflects hepatic and, to a lesser extent, cardiac or muscle integrity.
Concentration of Total Serum Bilirubin Measured by Diazo Method (mg/dL) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Total bilirubin will be measured using a diazo-based colorimetric assay and expressed in milligrams per deciliter (mg/dL). Bilirubin serves as an indicator of liver function and hemolysis.
Concentration of High-Sensitivity C-Reactive Protein (hs-CRP) Measured by Immunoturbidimetric Assay (mg/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  High-sensitivity C-reactive protein will be measured using an immunoturbidimetric assay and expressed in milligrams per liter (mg/L). hs-CRP serves as a marker of systemic inflammation and cardiovascular risk.
Concentration of Asymmetric Dimethylarginine (ADMA) Measured by Liquid Chromatography-Tandem Mass Spectrometry (µmol/L) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Asymmetric dimethylarginine (ADMA) will be quantified using LC-MS/MS and expressed in micromoles per liter (µmol/L). ADMA reflects endothelial function and nitric oxide metabolism.
Concentration of Platelet Factor 4 (PF4) Measured by Enzyme-Linked Immunosorbent Assay (ng/mL or OD Units) | Measured 1 month before, 7 days before, and then 3 days, 7 days, 1 month, 3 months, and 6 months after treatment.
  Platelet Factor 4 (PF4) will be measured using a validated ELISA. Results will be reported as nanograms per milliliter (ng/mL) or optical density (OD) units, depending on assay type. PF4 is a marker of platelet activation and potential immune-mediated coagulation effects.
Epigenetic Biological Age Estimated From Whole-Genome DNA Methylation Profiles (years) | Measured 7 days before administration and then 3 days, 7 days, 1 month, 3 months, and 6 months after administration
  Whole-blood DNA methylation will be measured using bisulfite sequencing performed by Generation Lab. Epigenetic biological age will be computed from these methylation data using validated algorithms. Age estimates will be expressed in years. Lower epigenetic age relative to chronological age indicates younger biological status.
Estimated Brain Age: Derived From Kernel Flow Functional Near-Infrared Spectroscopy (fNIRS) Analysis (years) | Measured 7 days before and then 3 days, 7 days, 1 month, and 3 months after treatment
  Resting-state cerebral hemodynamic activity will be measured using the Kernel Flow headset, which integrates time-domain functional near-infrared spectroscopy (TD-fNIRS) and behavioral data. Kernel's proprietary machine learning algorithms will process whole-brain optical signals to generate an Estimated Brain Age, expressed in years. The metric represents the predicted biological brain age relative to chronological age, derived from composite models trained on resting-state fNIRS and behavioral features. Lower Estimated Brain Age values indicate more youthful brain function. Data will be reported per participant at baseline and after treatment.
Cognitive Performance Index and Domain Percentiles Derived From Kernel Flow functional near-infrared spectroscopy (fNIRS) and Behavioral Metrics (percentile where higher = better) | Measured 7 days before and then 3 days, 7 days, 1 month, and 3 months after treatment
  Cognitive performance will be assessed using Kernel Flow's composite metrics derived from time-domain functional near-infrared spectroscopy (TD-fNIRS) and brief behavioral tasks. Domain-specific percentile scores will be generated for Complex Attention, Executive Function, Learning and Memory, Language, and Perceptual-Motor Control, as well as an overall Cognitive Performance Index. Each score reflects age-normed percentile performance, integrating brain and behavioral features using Kernel's proprietary machine learning models. Higher percentiles indicate better cognitive performance relative to age-matched norms. Metrics will be reported per participant at baseline and after treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Apeiron Center, Austin, Texas, United States
- GARM Clinic, Roatán, Bay Islands, Honduras

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available along with a data dictionary describing each variable. If the study results in multiple publications, the IPD corresponding to the measures reported in each publication will be shared upon that publication. The complete trial dataset, if anything is remaining, will be made available once all results have been published. Supporting documentation shared will include study protocol, statistical analysis plan, informed consent forms, and analytic code.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available upon publication and will be available indefinitely.
Access Criteria: Data will be made available to anyone who wishes to access it in an online repository at Vivli (https://vivli.org/). The types of data shared will include de-identified data of pre- and post-treatment values for the following measures: serum Klotho levels; kidney and blood safety panels; questionnaires and adverse event reporting data (all check box questions; however, any open-ended answer data will reviewed to ensure they cannot be used to identify an individual participant - final judgments will be made by the study central coordinator); RIAS-2 scores; all NIH-toolbox measures; Kernel brain data; epigenetic age.

REFERENCES:
- [Background] Urakawa I, Yamazaki Y, Shimada T, Iijima K, Hasegawa H, Okawa K, Fujita T, Fukumoto S, Yamashita T. Klotho converts canonical FGF receptor into a specific receptor for FGF23. Nature. 2006 Dec 7;444(7120):770-4. doi: 10.1038/nature05315. Epub 2006 Oct 29. PMID 17086194
- [Background] Matsumura Y, Aizawa H, Shiraki-Iida T, Nagai R, Kuro-o M, Nabeshima Y. Identification of the human klotho gene and its two transcripts encoding membrane and secreted klotho protein. Biochem Biophys Res Commun. 1998 Jan 26;242(3):626-30. doi: 10.1006/bbrc.1997.8019. PMID 9464267
- [Background] Masso A, Sanchez A, Bosch A, Gimenez-Llort L, Chillon M. Secreted alphaKlotho isoform protects against age-dependent memory deficits. Mol Psychiatry. 2018 Sep;23(9):1937-1947. doi: 10.1038/mp.2017.211. Epub 2017 Oct 31. PMID 29086766
- [Background] Masso A, Sanchez A, Gimenez-Llort L, Lizcano JM, Canete M, Garcia B, Torres-Lista V, Puig M, Bosch A, Chillon M. Secreted and Transmembrane alphaKlotho Isoforms Have Different Spatio-Temporal Profiles in the Brain during Aging and Alzheimer's Disease Progression. PLoS One. 2015 Nov 24;10(11):e0143623. doi: 10.1371/journal.pone.0143623. eCollection 2015. PMID 26599613
- [Background] Imura A, Tsuji Y, Murata M, Maeda R, Kubota K, Iwano A, Obuse C, Togashi K, Tominaga M, Kita N, Tomiyama K, Iijima J, Nabeshima Y, Fujioka M, Asato R, Tanaka S, Kojima K, Ito J, Nozaki K, Hashimoto N, Ito T, Nishio T, Uchiyama T, Fujimori T, Nabeshima Y. alpha-Klotho as a regulator of calcium homeostasis. Science. 2007 Jun 15;316(5831):1615-8. doi: 10.1126/science.1135901. PMID 17569864
- [Background] Kuro-o M, Matsumura Y, Aizawa H, Kawaguchi H, Suga T, Utsugi T, Ohyama Y, Kurabayashi M, Kaname T, Kume E, Iwasaki H, Iida A, Shiraki-Iida T, Nishikawa S, Nagai R, Nabeshima YI. Mutation of the mouse klotho gene leads to a syndrome resembling ageing. Nature. 1997 Nov 6;390(6655):45-51. doi: 10.1038/36285. PMID 9363890
- [Background] Imura A, Iwano A, Tohyama O, Tsuji Y, Nozaki K, Hashimoto N, Fujimori T, Nabeshima Y. Secreted Klotho protein in sera and CSF: implication for post-translational cleavage in release of Klotho protein from cell membrane. FEBS Lett. 2004 May 7;565(1-3):143-7. doi: 10.1016/j.febslet.2004.03.090. PMID 15135068
- [Background] Gupta S, Moreno AJ, Wang D, Leon J, Chen C, Hahn O, Poon Y, Greenberg K, David N, Wyss-Coray T, Raftery D, Promislow DEL, Dubal DB. KL1 Domain of Longevity Factor Klotho Mimics the Metabolome of Cognitive Stimulation and Enhances Cognition in Young and Aging Mice. J Neurosci. 2022 May 11;42(19):4016-4025. doi: 10.1523/JNEUROSCI.2458-21.2022. Epub 2022 Apr 15. PMID 35428698
- [Background] Dubal DB, Yokoyama JS, Zhu L, Broestl L, Worden K, Wang D, Sturm VE, Kim D, Klein E, Yu GQ, Ho K, Eilertson KE, Yu L, Kuro-o M, De Jager PL, Coppola G, Small GW, Bennett DA, Kramer JH, Abraham CR, Miller BL, Mucke L. Life extension factor klotho enhances cognition. Cell Rep. 2014 May 22;7(4):1065-76. doi: 10.1016/j.celrep.2014.03.076. Epub 2014 May 10. PMID 24813892
- [Background] Davidsohn N, Pezone M, Vernet A, Graveline A, Oliver D, Slomovic S, Punthambaker S, Sun X, Liao R, Bonventre JV, Church GM. A single combination gene therapy treats multiple age-related diseases. Proc Natl Acad Sci U S A. 2019 Nov 19;116(47):23505-23511. doi: 10.1073/pnas.1910073116. Epub 2019 Nov 4. PMID 31685628
- [Background] Chen CD, Podvin S, Gillespie E, Leeman SE, Abraham CR. Insulin stimulates the cleavage and release of the extracellular domain of Klotho by ADAM10 and ADAM17. Proc Natl Acad Sci U S A. 2007 Dec 11;104(50):19796-801. doi: 10.1073/pnas.0709805104. Epub 2007 Dec 3. PMID 18056631
- [Background] Castner SA, Gupta S, Wang D, Moreno AJ, Park C, Chen C, Poon Y, Groen A, Greenberg K, David N, Boone T, Baxter MG, Williams GV, Dubal DB. Longevity factor klotho enhances cognition in aged nonhuman primates. Nat Aging. 2023 Aug;3(8):931-937. doi: 10.1038/s43587-023-00441-x. Epub 2023 Jul 3. PMID 37400721
- [Background] Arking DE, Krebsova A, Macek M Sr, Macek M Jr, Arking A, Mian IS, Fried L, Hamosh A, Dey S, McIntosh I, Dietz HC. Association of human aging with a functional variant of klotho. Proc Natl Acad Sci U S A. 2002 Jan 22;99(2):856-61. doi: 10.1073/pnas.022484299. Epub 2002 Jan 15. PMID 11792841
- [Background] Abraham CR, Mullen PC, Tucker-Zhou T, Chen CD, Zeldich E. Klotho Is a Neuroprotective and Cognition-Enhancing Protein. Vitam Horm. 2016;101:215-38. doi: 10.1016/bs.vh.2016.02.004. Epub 2016 Mar 22. PMID 27125744